CLINICAL TRIAL: NCT00582816
Title: Reduced Intensity Haploidentical Transplantation With NK Cell Infusion for Pediatric Acute Leukemia and High Risk Solid Tumors, BMT06407
Brief Title: Haploidentical Transplant With NK Cell Infusion for Pediatric Acute Leukemia and Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: toxicity
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT06407; H-2006-0297 (Other: UW IRB); 2012-0661 (Other: UW IRB); A536700 (Other: UW Madison); SMPH\PEDIATRICS\PEDIATRICS (Other: UW Madison); NCI-2011-00687 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-07

CONDITIONS: Leukemia; Solid Tumors
Keywords: Recurrent or Refractory Leukemia or Solid Tumors in Pediatrics
MeSH Terms: conditions — Leukemia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): patients will undergo a standard pre-transplant evaluation, but will also have blood drawn to evaluate their HLA class I killer immunoglobulin-like receptor (KIR) ligand typing. Parents will undergo KIR genotyping and phenotyping, and a donor will be selected based on which parent shows the greatest degree of KIR receptor-ligand mismatching. Once the donor has been selected he/she will undergo a peripheral blood stem cell (PBSC) collection utilizing G-CSF and GM-CSF for stem cell mobilization. The PBSC collection will be performed utilizing standard procedures. The PBSC will then be processed in the UW BMT Laboratory in order to deplete the graft of T cells. This will be accomplished using the CliniMACS cell separation system. T cell depletion is a standard procedure for patients receiving haploidentical stem cell grafts. The resulting stem cell product will be analyzed for T cell, stem cell and NK cell content.
  Interventions: Device: Clinimacs Cell Separation System; Drug: conditioning chemotherapy; Other: DLI

INTERVENTIONS:
Device: Clinimacs Cell Separation System — Depletion of T-cells
Drug: conditioning chemotherapy — Methylprednisolone, Equine ATG, Cyclosporine, Fludarabine, Melphalan, Thiotepa and Rituximab.
Other: DLI — NK Cell selected DLI

SUMMARY:
This study will assess the feasibility of utilizing a reduced intensity conditioning regimen, in the setting of haploidentical transplantation, for patients with recurrent acute lymphoblastic leukemia (ALL), AML and high risk or refractory solid tumors. In addition, the feasibility and safety of administering post-transplant NK cell infusions will be evaluated. Data obtained from this study will help determine the efficacy of allogeneic HSCT in the treatment of pediatric sarcomas and add to the small body of literature utilizing haploidentical HSCT to treat acute leukemia in pediatric patients. This study will also further elucidate the role of NK cells in mediating a graft vs. tumor effect in allogeneic HSCT. The main benefit to society is that this study will explore a novel therapy for children with highly refractory cancer who are felt to be incurable with conventional approaches. If feasibility is demonstrated, and there is evidence of anti-tumor activity, then this will open up a new area of clinical research to better define the efficacy of this approach for specific childhood malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumors that have failed auto transplant or are ineligible to receive auto transplant
* Relapsed AML in 1st relapse or 2nd or 3rd CR
* Relapsed ALL if they fail to attain an initial remission or if they relapse within 1 year following the discontinuation of chemotherapy.
* Greater than or equal to 6 months and <26 years old
* Suitable haploidentical donor available

Exclusion Criteria:

* Leukemia with >25% blasts in bone marrow at the time of admission to the HSCT unit.
* Serum bilirubin >3 mg/dl
* GFR <40 ml/min/1.73 mw
* Cardiac left ventricular ejection fraction <40%
* HIV+
* Pregnant

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth DeSantes, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Kenneth DeSantes., MD, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with relapsed acute leukemia and very high-risk solid tumors. The last subject was enrolled in October 2013.
Groups:
- Haploidentical Transplant With NK Cell Infusion: Patients underwent a standard pre-transplant evaluation, but will also had blood drawn to evaluate their HLA class I killer immunoglobulin-like receptor (KIR) ligand typing. Parents underwent KIR genotyping and phenotyping, and a donor was selected based on which parent showed the greatest degree of KIR receptor-ligand mismatching. When the donor had been selected he/she underwent a peripheral blood stem cell (PBSC) collection utilizing G-CSF and GM-CSF for stem cell mobilization. The PBSC collection was performed utilizing standard procedures. The PBSC was then be processed in the UW BMT Laboratory in order to deplete the graft of T cells. This was accomplished using the CliniMACS cell separation system. T cell depletion is a standard procedure for patients receiving haploidentical stem cell grafts. The resulting stem cell product were analyzed for T cell, stem cell and NK cell content.
  Clinimacs Cell Separation System: Depletion of T-cells
Period: Overall Study
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Started | 9
Completed | 6 ("Completed" here means patients stably engrafted with donor cells.)
Not Completed | 3
Not completed — Engraftment Failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Grade III or IV GVHD
Description: Skin Grade III: Stage 0-4 GVHD, where 0 is no rash and 4 is generalized erythroderma with bullous formation and/or with desquamation Grade IV: Stage 4 GVHD, generalized erythroderma with bullous formation and/or with desquamation
  GI (diarrhea) Grade III: Stage 2-4 GVHD, where 2 is > 1000 mL/day but ≤ 1500 mL/day or 556-833 mL/m2, and 4 is severe abdominal pain +/- ileus or stool with frank blood or melena Grade IV: Stage 0-4 GVHD, where 0 is < 500 mL/day or 280 mL/m2, and 4 is severe abdominal pain +/- ileus or stool with frank blood or melena
  Overall:
  Grade III: Grade III Skin and/or GI as well as bilirubin 3.1-15 mg/dl Grade IV: Grade IV Skin and/or GI as well as bilirubin > 15 mg/dl
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 9
participants
  Grade III GVHD - Skin | 3
  Grade IV GVHD - GI | 2
  Grade III GVHD - GI | 1
  Overall Grade III GVHD | 2
  Overall Grade IV GVHD | 2

2. Primary Outcome: Engraftment Failure
Description: Utilize non-myeloablative conditioning regimen in the haploidentical transplant setting.
  Primary engraftment failure: failure to achieve ANC of ≥500/uL prior to day +28 Late engraftment failure: Initial engraftment achieved with ANC ≥500/uL by day +28 followed by loss of graft Autologous Cells Infused: achieved hematologic recovery following infusions of autologous stem cells Second Haploidentical Transplant: re-transplantation utilizing an alternative haploidentical donor
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 9
participants
  Primary Engraftment Failure | 2
  Late Engraftment Failure | 1
  Autologous Cells Infused | 2
  Second Haploidentical Transplant | 1

3. Primary Outcome: Number of Days Until Engraftment Criteria Were Met
Description: Utilize non-myeloablative conditioning regimen in the haploidentical transplant setting. Engraftment is defined as achieving an absolute neutrophil count ≥ 500 by 28 days post-transplant; platelets and red blood cells will also be measured up to 28 days:
  * Neutrophils: ≥500/uL for 3 days
  * Platelets: ≥20 K/uL for 3 days without transfusion
  * Red blood cells: the date of the last RBC transfusion after achieving transfusion independence Results are reported as number of days until engraftment criteria was met, per neutrophil, platelet and red blood cell measurements, above.
Time Frame: 28 days
Measure: Median (Full Range); unit: days
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 7
days
  Neutrophils | 18 [14 to 20]
  Platelets | 16 [10 to 21]
  Red Blood Cells | 16 [8 to 22]

4. Primary Outcome: Mortality Rate
Description: Mortality rate at 100 days post-transplant.
Time Frame: 100 days post-transplant
Population: Death Prior to Day +100
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 9
participants | 1

5. Secondary Outcome: NK Expression Levels
Description: Natural Killer (NK) cell expression levels will be explored. Blood samples will be collected at months 1, 2, 3, 6, 9, and 12.
Time Frame: Up to 12 months
Population: Blood samples were not collected uniformly as many patients developed GVHD, requiring treatment with steroids. Once steroids were initiated the results of this testing became uninterpretable. No data was collected towards this outcome measure.
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 0

6. Secondary Outcome: Association Between Parental KIR Genotypes and NK Cell Cytotoxicities
Description: NK cells express killer-cell immunoglobulin-like receptors (KIR) and have cytotoxic activity. The association between NK cell cytotoxicity over time and KIR genotypes will be examined. Blood samples will be collected at months 1, 2, 3, 6, 9, and 12.
Time Frame: Day 60
Population: as for outcome 5
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 0

7. Secondary Outcome: Analysis of NK Cell KIR Expression Over Time
Description: NK cell KIR expression over time will be examined. Blood samples will be collected at months 1, 2, 3, 6, 9, and 12.
Time Frame: Up to 12 months
Population: as for outcome 5
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 3 years.
Description: Adverse events were routinely determined to have occurred by regular investigator assessment and regular laboratory testing.
Arm/Group | Haploidentical Transplant With NK Cell Infusion
Serious Adverse Events (participants affected / at risk) | 8/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Transplant With NK Cell Infusion (N=9)
Grade 3 infection (Infections and infestations) | 4 (5)
Grade 3 anorexia (Metabolism and nutrition disorders) | 3 (3)
Grade 3 diarrhea (Gastrointestinal disorders) | 2 (2)
Grade 3 GVHD (Blood and lymphatic system disorders) | 2 (2)
Grade 2 seizure (Nervous system disorders) | 2 (2)
Grade 4 engraftment failure possibly from CMV riemia or inadequate stem cell dose (Blood and lymphatic system disorders) | 1 (1)
Grade 4 engraftment failure (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 1 (1)
Grade 3 dehydration (Metabolism and nutrition disorders) | 1 (1)
Grade 2 diarrhea (Gastrointestinal disorders) | 1 (1)
Grade 1 fever (General disorders) | 1 (1)
Grade 3 fever (General disorders) | 1 (1)
Grade 2 acute GVHD (Blood and lymphatic system disorders) | 1 (1)
Grade 3 skin GVHD (Skin and subcutaneous tissue disorders) | 1 (1)
Grade 4 graft rejection (Blood and lymphatic system disorders) | 1 (1)
Grade 3 hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Grade 4 infection (Infections and infestations) | 1 (1)
Grade 1 leukoencephalopathy (Nervous system disorders) | 1 (1)
Grade 2 pain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study involved a small patient cohort; blood samples were to be collected towards the secondary outcome measures. Unfortunately, participants whose blood samples were collected developed GVHD and the tests became uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No